CLINICAL TRIAL: NCT03243318
Title: Motor Evoked Potential in the Affected Upper Limb Predicts the Potential of Motor Recovery in Subacute Stroke Patients
Status: Completed | Type: Observational
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Eric Man Pun Yeung, Doctor, Hospital Authority, Hong Kong
Other Study IDs: KHMEPsUL2017
Record Dates: First submitted 2017-08-04; First posted 2017-08-09 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Stroke, Subacute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Presence of motor evoked potentials: Those patients with Shoulder Abduction and Finger Extension (SAFE) score <8/10 with the presence of motor evoked potentials elicited by TMS over the ipsilesional motor cortex
  Interventions: Diagnostic Test: MEPs induced by TMS
- absence of motor evoked potentials: Those patients with Shoulder Abduction and Finger Extension (SAFE) score <8/10 with the absence of motor evoked potentials elicited by TMS over the ipsilesional motor cortex
  Interventions: Diagnostic Test: MEPs induced by TMS

INTERVENTIONS:
Diagnostic Test: MEPs induced by TMS — Using TMS induced MEPs over motor cortex of the affected side to predict motor recovery potentials

SUMMARY:
Stroke is the third common cause of adult disability in dveloped countries. Early identification of the potential for motor recovery is important to avoid 'learned disuse' and to initiate appropriate therapy with achievable goals. The current cohort study focuses on those patients with SAFE <8 and using motor evoked potentials (MEPs) to improve on prognostication of upper limb motor recovery among subacute stroke patients in a local stroke population.

ELIGIBILITY:
Inclusion Criteria:

* First stroke with hemiparesis or hemiplegia with SAFE <8

Exclusion Criteria:

* contra-indication to TMS or MRI, history of seizure, pregnancy and mentally unfit to understand the consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subacute stroke patients
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test | Change of Baseline Action Research Arm Test at 12 weeks post-stroke
  Upper limb functional test

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation, Kowloon Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No